CLINICAL TRIAL: NCT01006460
Title: A Randomized, Placebo Controlled, Parallel, Double Blinded Trial With Rhodiola Rosea Extract SHR-5 (Arctic Root) Compared With the Extract When Combined With Schizandra and Russian Root (Adapt 232), Standardized Ginseng Extract and Placebo Regarding Impact on the Level of Energy, Ability to Work Under Stress, Quality of Life and Wellbeing, in Middleaged Women Who Are Still Employed
Brief Title: A Study With Arctic Root Compared With the Extract When Combined With Schizandra and Russian Root (Adapt 232), Standardized Ginseng Extract and Placebo Regarding Impact on the Level of Energy, Ability to Work Under Stress, Quality of Life and Wellbeing, in Middleaged Women Who Are Still Employed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Kaj Winther Hansen, Frederiksbegg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR5/DK
Record Dates: First submitted 2009-11-01; First posted 2009-11-02 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2009-11

CONDITIONS: Depression; Stress
Keywords: Quality of life and subjective well-being in middle aged women
MeSH Terms: conditions — Depression | interventions — Siberian ginseng root; schizandrin; Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Adapt 232 (Experimental)
  Interventions: Drug: Rhodiola rosea, L., Eleutherococcus senticosus, Schisandra chinensis
- Arctic root group (Experimental)
  Interventions: Drug: Rhodiola rosea, L
- Ginseng group (Active Comparator)
  Interventions: Drug: Panax ginseng
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo - dark brown sugar

INTERVENTIONS:
Drug: Rhodiola rosea, L — 3 Capsules twice a day
  Arms: Arctic root group
Drug: Rhodiola rosea, L., Eleutherococcus senticosus, Schisandra chinensis — 3 capsules twice a day
  Arms: Adapt 232
Drug: Panax ginseng — 3 capsules twice a day
  Arms: Ginseng group
Drug: Placebo - dark brown sugar — 3 capsules twice a day
  Arms: Placebo group

SUMMARY:
This is clinical trial to document the efficacy of a proprietary standardized extract of Arctic root in comparison to a standardized commercial extract of ginseng and placebo from an every day consumer perspective to ameliorate mild depression, reduce stress and improve quality of life. A newly developed adaptogenic formulation, Adapt 232, was included into the study in order to evaluate its effect in comparison to the others.

ELIGIBILITY:
Inclusion Criteria:

* healthy females, over 40 years of age, who have stated that they for a longer period of time have felt stressed due to demanding daily activities at work and/or at home.

Exclusion Criteria:

* suffering from any known medical disease, e.g. cardiovascular, joint, and liver or kidney diseases, cancer, or psychiatric disease.
* with a psychiatric diagnose, using narcotics or suffering from HIV.
* with known allergy to any of the study medications.
* misusing euphorizing or pain killing drugs
* having used any adaptogenic product the last 2 months.
* having used cortisol or any other corticosteroid products the last 6 months
* being pregnant or breast-feeding
* which at the first interview are judged to be not cooperative or not to be able to finalize the study

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Psychological parameters: changes in cognitive functions as measured by the D2 Test of Attention | Over a period of 28 days of treatment

SECONDARY OUTCOMES:
Depression parameters: changes in depressive state as measured by the using Hamilton Depression Rating Scale (HAM-D) and Bechs Depression Inventory (BDI). | over a period of 28 days of treatment
Quality of Life parameters: changes in quality of life as measured by the SF-36 scale, Danish Stress Profile (SP) test and questions regarding various aspects of well-being as formulated in a non-validated VAS scale | Over a period of 28 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kaj Winther, Dr, Principal Investigator — Clinical Biochemistry department, Frederiksberg Hospital
Locations (1):
- Department of Clinical Biochemistry, Frederikbergs Hospital, Frederiksberg, Denmark